CLINICAL TRIAL: NCT01390103
Title: Do Hip Injections Improve Short-Term Biomechanical Outcomes In Patients With Hip Pain
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 711-2010
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Hip Pain
Keywords: hip pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Assessment following the hip injection: Assessment to evaluate the effect of the hip injection on biomechanics.
  Interventions: Other: Assessment following hip injection

INTERVENTIONS:
Other: Assessment following hip injection — Assessment to evaluate the effect of the hip injection on biomechanics.

SUMMARY:
The purpose of this project is to determine the effect of hip injections on hip biomechanics in patients with hip pain.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis patients with hip pain requiring hip injection
* Receiving hip injection
* BMI < 35

Exclusion Criteria:

* BMI > 35
* severely impaired intellectual capacity
* dementia, or other neurodegenerative diseases that would preclude appropriate cognitive or physical ability to perform study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be all patients receiving a hip injection for hip pain.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Determine the immediate biomechanical effect in patients that receive a hip injection. | The short-term biomechanical effects of the hip will be evaluated within 1 hour of the patient receiving the injection.
  The biomechanical assessment of gait will consist of walking on a gait mat. The mat is a specialized pressure sensor system. Prior to data collection, each participant will walk across the mat three times for acclimation. The first assessment will include a walk at a self-selected, comfortable pace across the mat, repeated three times. The second assessment will include walking as quickly as possible, also repeated three times.

SECONDARY OUTCOMES:
Oswestry Hip Pain Disability Questionnaire | Baseline, Within 1 hour of hip injection, 2 weeks post-injection
  Oswestry Hip Pain Disability Questionnaire. This a standard, well validated questionnaire to assess disability caused by hip pain. The questionnaire is a 10-item scale, ranging from 0 to 100%, to obtain a score for functional disability caused by hip pain.
Medical Outcomes Study (MOS) Short-Form Health Survey (SF-12) | Baseline, Within 1 hour of injection, 2 weeks post-injection
  The SF-12 is a global health assessment questionnaire ranging from 0 to 100%, to score self-experienced health related to quality of life. Items are grouped into two domains from which an overall summary score, a physical component score and a mental component score can be derived. A high score on each of the scales reflects a high level of self-experienced health
10 centimeter Visual Analog Scale (VAS) | Baseline, Within 1 hour of injection, 2 weeks post-injection
  Hip pain is a symptom that affects the overall Quality Of Life. Hip pain intensity will be self-assessed by a 10 cm visual analogue scale with terminal descriptors (anchors of 0 cm = no pain; 10 cm = worst possible pain). The VAS is an accepted outcome measure for chronic pain conditions.
Pain Provocative Maneuvers | Baseline, Within 1 hour of injection, 2 weeks pos-injection
  All patients currently undergoing hip injections receive a basic physical exam including patient specific provocative maneuvers both before and after the injection. The loss of pain after injection of a local anesthetic is part of the routine treatment algorithm and the results will be correlated with other outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: MaryBeth Horodyski, PhD, Study Director — University of Florida Departmen of Orthopaedics
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States